CLINICAL TRIAL: NCT06834958
Title: Clinical Diagnosis of Acute Appendicitis with Normal WBCS Count with Role of Inflammatory Markers and Radiology
Status: Active, not recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrhman Kotb, Surgeon, Assiut University
Other Study IDs: Clinical diagnosis of acute ap
Record Dates: First submitted 2025-01-31; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Acute Appendicitis
Keywords: Clinical diagnosis of acute appendicitis
MeSH Terms: conditions — Appendicitis | interventions — Appendectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patient included who have acute appendicitis clinically and normal WBCS count
  Interventions: Procedure: Appendectomy

INTERVENTIONS:
Procedure: Appendectomy — Open surgery for appendix which is inflamed

SUMMARY:
The aim of this study is to describe the proportion of pa-tients with normal preoperative inflammatorymarkers among patients with histopathologically proven acute appendicitis

DETAILED DESCRIPTION:
2.4.1- Type of the study: prospective clinical trial study 2.4. 2- Study Setting: Assuit university hospital 2.4. 3- Study subjects:

1. Inclusion criteria:

   patients complain of Rt iliac pain with Us positive for acute appendicitis with WBCS normal .
2. Exclusion criteria:

malignant mass cancer appendix mesenteric adentis cecal diverticulum salpingitis c. Sample Size Calculation: 50 cases 2.4.4 -Study tools (in detail, e.g., lab methods, instruments, steps, chemicals, …): Lab WBCS count CRP level Neutrophil differential count Clinical correlation US findings and MSCT if needed

ELIGIBILITY:
Inclusion

* Male or female patients é clinically diagnosed acute appendicitis with normal WBCS

Exclusion Criteria:

* complicated AA (perforation, peri appendicular abscess or suspicion of a tumor.

  2_inflammatory bowel diseases 3_inability to co-operate and give informed consent 4_diffuse peritonitis 5_Patients with serious comorbid conditions DM & renal insufficiency, serum creatinine > 150 μmol/l 6_Pregnant & lactating patient 7_Patients with advanced malignancies & pt on immunosuppressive drugs

Ages: 14 Days to 60 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Study not need special type of people
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Surgery done if needed | Days of hospital reservation
  Patient with acute appendicitis and normal WBCS count will be under observation for while but people with evidence on imaging and high inflammatory markers will go under surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Assuit university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- See also: Related Info — https://www.ncbi.nlm.nih.gov/books/NBK493193/